CLINICAL TRIAL: NCT00473122
Title: Delayed-Immediate Breast Reconstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0955; NCI-2012-02091 (Registry Identifier: NCI CTRP); BCTR0503938 (Other: Susan G. Komen Breast Cancer Foundation)
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Reconstruction; Delayed-Immediate Reconstruction; Postmastectomy Radiation Therapy; Mastectomy; XRT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Delayed-Immediate Breast Reconstruction (Other): Delayed-Immediate Reconstruction: If radiation therapy (XRT) not needed, immediate reconstruction. If XRT is needed, delayed reconstruction until XRT complete.
  Interventions: Procedure: Delayed-Immediate Breast Reconstruction

INTERVENTIONS:
Procedure: Delayed-Immediate Breast Reconstruction — Immediate reconstruction surgery if no XRT required; or reconstruction surgery delayed until XRT complete.

SUMMARY:
The goal of this clinical research study is to evaluate a new two-stage approach (delayed-immediate reconstruction) to breast reconstruction in women who may require post-mastectomy radiation therapy. Researchers will compare the cosmetic outcomes and any complications that occur in women who receive delayed-immediate reconstruction to those who receive the standard approaches (either immediate reconstruction or delayed breast reconstruction).

DETAILED DESCRIPTION:
In women who have a mastectomy and desire breast reconstruction, the best timing of breast reconstruction depends on whether radiation therapy (XRT) is needed. If XRT is not needed, immediate reconstruction offers the best cosmetic result. However, if XRT is needed, it is better to delay reconstruction until XRT is complete. There are 2 reasons to wait. First, the presence of a reconstructed breast can interfere with the delivery of XRT, decreasing the effectiveness of this treatment. Second, exposing a reconstructed breast to radiation can cause poor cosmetic results. Today, many women are not offered immediate reconstruction because it is not known at the time of their mastectomy whether they will need XRT. Researchers believe that for such women, a new approach called "delayed-immediate reconstruction" will offer the cosmetic benefits of immediate reconstruction without the potential drawbacks of ineffective treatment.

If you agree to take part in this study, you will have your already scheduled skin-sparing mastectomy. However, at the time of your routine mastectomy, you will also have a tissue expander or postoperatively adjustable implant (fully inflated with saline or as allowed by the remaining capacity [space] of the retained breast skin) placed in your breast. Some patients will have a small biopsy of skin, that is normally discarded, done so that scientists can learn about changes and ways of healing after radiation. When the final pathology report is complete (about 1 week after mastectomy), the radiation doctor and/or your surgeon will decide whether or not you need XRT.

If the results show that you do not need XRT, you will have the tissue expander or implant removed and will have standard definitive breast reconstruction, using the preserved breast skin about 2 weeks after mastectomy. The reconstructive technique used will be decided based on anatomical considerations, surgical factors, and your personal desires. The postoperative follow-up will be similar to that of patients who have standard immediate breast reconstruction.

If the results show that you do need XRT, the tissue expander or adjustable implant will be completely deflated in the plastic surgery clinic before you receive standard XRT. Radiation must be given either at MD Anderson or an MD Anderson-affiliated site. Deflation of the tissue expander or implant will result in a flat chest wall that will decrease difficulties with radiation delivery that can occur after an immediate breast reconstruction. If you also require chemotherapy after mastectomy, the tissue expander or implant will remain inflated during chemotherapy (additional saline-filling may also be performed during chemotherapy, if required). In patients who have already received chemotherapy before mastectomy or who will not require chemotherapy, the expander or implant will remain inflated during the 4-to-6-week period between mastectomy and XRT. About 3 weeks into your radiation treatments, you will come in to the plastic surgery clinic for a follow-up to check on the status of the implants.

Several weeks after the completion of XRT, the tissue expander or postoperatively adjustable implant will be gradually re-expanded over about 6-months. The internal scar capsule that forms around the tissue expander or implant before deflation usually allows for re-expansion after radiation therapy. Re-expansion after radiation therapy will be performed during postoperative visits to the plastic surgery clinic every 2-to-4 weeks until the desired size is achieved. About 6 months after the completion of XRT, a "skin-preserving" delayed reconstruction with a preference for autologous tissues only (no breast implants) will be performed. This will involve removal of the tissue expander or implant and definitive breast reconstruction. At the time of the skin-preserving delayed reconstruction, a small biopsy of usually thrown away radiated breast tissue as well as a sample of the skin, that is normally discarded, of the flap (your tissue that is taken from your back, stomach or buttock to build the breast) and a sample of the implant or tissue expander will be collected for laboratory evaluation. Researchers will evaluate the skin changes from radiation and expansion as well as from the internal scar capsule. This will be compared to radiated skin biopsies without expansion and biopsies taken after skin expansion without radiation.

Your medical information and photographs of your breast(s) will be gathered throughout the various stages of delayed-immediate reconstruction.

Delayed-immediate breast reconstruction is a two-stage approach and as such involves at least 2 surgical procedures. This does not include the possibility of procedures needed to modify the reconstructed breast, a procedure on the healthy breast to make it symmetrical (similar in appearance and size) with the reconstructed breast, and any nipple reconstruction and areolar tattooing that may be needed. If, later on, it is necessary to revise the reconstructed breast, a small skin sample (smaller than a pencil eraser) will again be collected for additional studies. This will not affect the outcome of your surgery or the way your breast will look.

The postoperative course, follow-up, and the need for additional surgical procedures will be decided in a similar fashion to that of standard immediate and delayed breast reconstruction.

This is an investigational study. The implants in this study have been FDA approved for skin expansion as a method of breast reconstruction. They are not specifically approved for both expansion and radiation. About 200 women will take part in this study. All will be enrolled at MD Anderson Cancer Center (MDACC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical stage I or stage II breast cancer who may require postmastectomy XRT.
2. Patients will be required to receive postmastectomy XRT as well as breast reconstructive procedures, including subsequent deflation and re-inflation of the prosthesis after XRT at University of Texas MD Anderson Cancer Center (UT MDACC).
3. Patients must sign the consent form and must be able to withstand two (2) anesthetic procedures.
4. Patients with stage I breast cancer who will be eligible for delayed-immediate breast reconstruction will have extensive microcalcifications within the affected by mammography that make it difficult to determine preoperatively the extent of invasive disease.

Exclusion Criteria:

1. Patients with stage III or stage IV breast cancer who are known preoperatively to require postmastectomy XRT.
2. Patients with stage I breast cancer who are unlikely to require postmastectomy XRT.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of Delayed-Immediate Breast Reconstruction | 5 Years
  Patient data and photographs gathered throughout the various stages of delayed-immediate reconstruction, during routine preoperative, intraoperative, and postoperative examinations. Details of primary disease include preoperative tumor stage, method of breast cancer diagnosis, tumor biologic characteristics, and the use of neoadjuvant chemotherapy. Preoperative and postoperative tumor stage compared to evaluate the indications for the delayed-immediate approach to breast reconstruction.

SECONDARY OUTCOMES:
Compare Aesthetic Outcomes for Immediate-Delayed Breast Reconstruction | 5 Years
  System used for aesthetic analysis is a four-point scale used to evaluate the aesthetic outcomes: excellent (4); good (3); fair (2); or poor (1). Results considered "excellent" when patient had almost perfect shape of the reconstructed breast and perfect contralateral breast symmetry, "good" when patient had imperfect shape of the reconstructed breast and imperfect contralateral symmetry but within normal limits, "fair" when patient had some contralateral asymmetry but a reasonably normal breast, and "poor" when patient had unacceptable shape and symmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Kronowitz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org